CLINICAL TRIAL: NCT02858349
Title: Mechanisms of Walking Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Pierce Boyne, Assistant Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-1916
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor was blinded to study design, including when participant was in control phase versus intervention phase
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 4-week control period with no intervention and 4-weeks of high-intensity interval training
  Interventions: Behavioral: No intervention; Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: No intervention — No intervention
Behavioral: High-intensity interval training — High-intensity walking exercise using bursts of concentrated effort alternated with recovery periods

SUMMARY:
Subjects with stroke will have behavioral testing and brain imaging before and after a 4-week control period and a 4-week exercise intervention.

DETAILED DESCRIPTION:
Subjects with stroke will have behavioral testing and brain imaging before and after a 4-week control period and a 4-week exercise intervention using high-intensity interval training.

ELIGIBILITY:
Inclusion Criteria:

* age 30-90 years
* unilateral stroke experienced >6 months prior to enrollment in middle cerebral artery (MCA) territory without complete disruption of the putamen on the lesion side
* walking speed <= 1.0 m/s on the 10 meter walk test
* able to walk 10m over ground with assistive devices as needed and no physical assistance

Exclusion Criteria:

* MRI incompatibility (e.g. metallic or electronic implants, severe claustrophobia)
* inability to perform mental imagery (time dependent motor imagery screening test [TDMI])
* evidence of significant arrhythmia or myocardial ischemia on treadmill ECG stress test, or significant baseline ECG abnormalities that would make an exercise ECG uninterpretable
* recent (<3 months) cardiopulmonary hospitalization
* unable to communicate with investigators or correctly answer consent comprehension questions
* significant ataxia or neglect (score of 2 on NIH stroke scale item 7 or 11)
* severe lower extremity (LE) spasticity (Ashworth >2)
* recent (<3 months) illicit drug or alcohol abuse or significant mental illness
* major post-stroke depression (PHQ-9 ≥10) in the absence of medical management
* participating in physical therapy or another interventional research study;
* recent (<3 months) paretic LE botulinum toxin injection
* concurrent progressive neurologic disorder or other major medical, orthopedic or peripheral vascular conditions that would limit improvement
* pregnancy

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Boyne, PT, DPT, NCS, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Comfortable Gait Speed, m/s [Mean (Standard Deviation); unit: meters per second] | 0.41 (0.33)
Stroke Chronicity [Mean (Standard Deviation); unit: years] | 2.4 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed
Description: 10-meter walk test
Time Frame: Change from 4-weeks to 8-weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second
Arm/Group | Arm 1
Number analyzed (Participants) | 10
meters per second | 0.13 [0.05 to 0.21]
Statistical Analysis 1: Comparison: Arm 1; Test type: Superiority; p = 0.0042, Mixed Models Analysis; Mean Difference (Net) = 0.13, 95% CI 2-sided [0.05 to 0.21]

2. Secondary Outcome: Gait Symmetry
Description: Paretic step ratio
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Metabolic Cost of Gait
Description: oxygen consumption rate during comfortable speed gait
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Aerobic Capacity
Description: oxygen consumption rate during exercise testing
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: NIH Toolbox - Cognition Domain
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: NIH Toolbox Standing Balance Test
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Stroke and Aphasia Quality of Life Scale
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Brain Locomotor Network Activation
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Brain Locomotor Network Connectivity
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Walking Capacity
Description: 6-minute walk test
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Daily Walking Activity
Description: activity monitor
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Walking Speed
Description: 10-meter walk test
Time Frame: baseline, 4 weeks, 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout study participation, which lasted approximately 4 months for each participant. The entire study lasted approximately 17 months.
Description: Each study visit, participant voluntary reporting of adverse events (AEs) was encouraged and AEs of interest were specifically queried, including: falls, orthopedic injuries, faintness, new/increased pain and muscle soreness. During clinical testing and training sessions, participants also had monitoring and post-session questioning to identify any signs or symptoms of cardiorespiratory insufficiency, new/worsening neurological impairments or orthopedic injury.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=10)
Dizziness (Nervous system disorders) | 4 (11)
Fall (Musculoskeletal and connective tissue disorders) | 5 (11)
Fatigue (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1) — Common cold
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased knee hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain/soreness (Musculoskeletal and connective tissue disorders) | 7 (24)
Surgical procedure (Musculoskeletal and connective tissue disorders) | 1 (1) — routine excision of ingrown toenail

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02858349/Prot_SAP_000.pdf